CLINICAL TRIAL: NCT06476912
Title: Investigating the Effects of Combined Balance Exercise and Vagus Nerve Stimulation on Weight-shifting Control and Ambulation in Patients With Parkinson Disease and Anxiety: Under Time and Space Constraints
Brief Title: Balance Exercise and Vagus Nerve Stimulation on Weight-shifting Control and Ambulation in Parkinson Disease and Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202301082RIND
Record Dates: First submitted 2024-05-03; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease
MeSH Terms: conditions — Parkinson Disease | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active VNS (Experimental): active vagus nerve stimulation
  Interventions: Other: weight-shifting exercise
- sham VNS (Sham Comparator): sham vagus nerve stimulation
  Interventions: Other: weight-shifting exercise

INTERVENTIONS:
Other: weight-shifting exercise — lateral weight-shifting balance training and VNS
  Other Names: vagus nerve stimulation

SUMMARY:
Postural balance and anxiety are the two critical factors for reducing independence and quality of life in patients with Parkinson's disease (PD). Anxiety would deteriorate balance and gait dysfunction. Especially, relative to non-constraint condition, PD patients with anxiety had greater increases in anxiety level and balance/gait impairment in time-constraint or space-constraint condition than PD patients without anxiety. Presently, the appropriate managements for reducing anxiety in patients with PD had not been comprehensively investigated. Vagus nerve stimulation (VNS) is one kind intervention of neuromodulation. Previous studies showed that VNS could reduce anxiety level for patients with anxiety syndrome. In addition, motor training with VNS could reinforce training benefits due to facilitation of brain plasticity. However, there is no study investigating the effect of VNS on anxiety in PD. Also, the effect of combined exercise training and VNS on balance and gait in PD has not been studied. With the use of behavior performance, skin conductance response, and electroencephalogram (EEG) measurement, the purpose of the 3-year research project is to investigate the effects of VNS on anxiety and balance/gait control in patients with PD. In the first year, we will investigate the immediate effect of VNS on anxiety and weight-shifting performance in conditions with time constraint and space constraint. In the second and third years, we will the investigate long-term effects of combined exercise training and VNS on anxiety level, weight-shifting and walking performance in time constraint condition and space constraint condition, respectively. The present project is expected to have significant contributions not only to gain a better insight to neural correlates of anxiety and balance control with VNS, but to optimize rehabilitation strategy for PD patients with anxiety.

DETAILED DESCRIPTION:
Anxiety is one of the most prevalent psychiatric comorbidities in patients with Parkinson disease (PD) and would deteriorate patients' motor symptom and quality of life. In particular, under space constraint condition, the increased anxiety level would impair balance control and ambulation in PD. Current pharmacological management and non-pharmacological management for reducing anxiety lack of significant efficacy. Vagus nerve stimulation (VNS) is a neurostimulation intervention for anxiety, and transcutaneous vagus nerve stimulation (tVNS) can be undergone with a transcutaneous electrical nerve stimulator, which is an accessible tool in clinic. However, there is no study investigating tVNS effects on anxiety reduction in PD. Therefore, the purpose of this study is to investigate the effect of combined balance training and tVNS on reducing anxiety and improving balance and gait in patients with PD, especially under space constraint condition.

ELIGIBILITY:
Inclusion Criteria:

1. idiopathic Parkinson's disease
2. Parkinson Anxiety Scale < 13 scores: non-anxiety group or PAS >14 scores: anxiety group
3. subject can walk for 20 meters without assistance
4. no other neurological disease

Exclusion Criteria:

1. Mini-Mental State Examination, MMSE < 26 scores
2. depression
3. brain surgery such as deep brain stimulation
4. people with visual impairments

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
EEG relative power | 10 minutes
  brain excitability

SECONDARY OUTCOMES:
Weight-shifting tracking error | 10 minutes
  behavior performance
Skin conductance level | 10 minutes
  sweat gland activation

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Ya Huang, PhD, Study Director — National Taiwan University
Locations (1):
- School and graduate institute of physical therapy, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to concerns about participant privacy and confidentiality. Although the data will be de-identified, we prioritize the protection of our participants' personal information.